CLINICAL TRIAL: NCT03029468
Title: A Three-arm Feasibility Study of Web- and Smartphone-delivered Cognitive Behavioral Therapy as an Adjunct to Opioid Pain Treatment Among Adults With Sickle Cell Disease (SCD)
Brief Title: Computerized Cognitive Behavioral Therapy Assisted Life Management for Pain in Sickle Cell Disease
Acronym: CALM-SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Toronto (Other); University of Washington (Other); Duke University (Other); Vanderbilt University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Charles Jonassaint, PhD, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO17010378; K23HL135396 (NIH)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Sickle Cell Disease; Chronic Pain
Keywords: Cognitive behavioral therapy; Chronic pain; Sickle cell disease; Mobile phone app; Mental health; Behavioral intervention; Behavioral health
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Three-arm feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computerized CBT (Experimental): Computerized cognitive behavioral therapy (cCBT) for pain via an integrated smartphone and web-based skills training program: The training plan will help users learn how to recognize negative thoughts and emotions, use cognitive skills and problem-solving, and apply coping behaviors such as distraction, activity scheduling, and relaxation. The cCBT arm emphasizes skills acquisition and learning through practice; thus, the program involves regular homework assignments, and follow-up with the care coach and social network about issues faced and what skills were or could be used. This intervention is consistent with the tailored behavioral services patients would receive individually or as a group when working with a psychologist or behavioral pain specialist.
  Interventions: Behavioral: cognitive behavioral therapy
- e-Education (Active Comparator): Participants will receive pain education through online modules that they will be asked to complete using their personal or study-provided smartphone. Each module includes learning tasks, a reading assignment, and a short quiz based on material. The education group will receive care coach contact on the same schedule as the cCBT group. The care coach will provide supportive therapy and encouragement to complete modules and apply the lessons to their daily life.
  Interventions: Behavioral: eEducation
- Usual Care (No Intervention): Participants who are not eligible or who are not randomized into one of the intervention arms of this study will serve as a comparison group to ensure we are treating a representative sample of patients. Further, patients who were eligible but were not randomized into one of the intervention arms will serve as a usual care control group.

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — CBT teaches users how to recognize negative thoughts and emotions, use cognitive skills and problem-solving, and apply coping behaviors such as distraction, activity scheduling, and relaxation.
  Arms: Computerized CBT
Behavioral: eEducation — Pain and sickle cell disease education delivered through a mobile electronic device
  Arms: e-Education

SUMMARY:
The primary aim of this study is to test the feasibility and acceptability of implementing a multimedia computerized cognitive behavioral therapy (cCBT) program for reducing SCD pain symptoms in a single-arm pilot pragmatic clinical trial. The investigators will recruit 40 SCD patients with chronic pain and/or on chronic opioid pain treatment and randomize them 3:1 to two groups (cCBT and e-Education respectively), randomizing unevenly in order to best gather feasibility data for the cCBT. Both groups will use a mobile app to track daily pain/mood. The cCBT group will receive sessions of the CALM-SCD program to complete via mobile device and will have weekly follow-up with a care coach. The Education group will receive online education modules to complete via mobile device and will also have weekly follow-up with a care coach. The primary outcomes of the trial include feasibility (recruitment, retention, provider and patient feedback) and acceptability (sessions completed) of the CALM-SCD program.

DETAILED DESCRIPTION:
The objective of this study is to provide the experiences and data that will support a later, larger, and adequately powered effectiveness trial of the CALM-SCD, computerized cognitive behavioral therapy (cCBT) program. The investigators hypothesize that CALM-SCD is acceptable, i.e., patients will use it (90% of users will complete the first lesson within 3 months; 70% will complete³4 sessions; 50% of users will complete all 8 sessions), and feasible, i.e., the investigators can recruit >80% of patients approached, and >90% of enrolled participants will complete their 6-month follow-up assessment. The investigators will also have preliminary data on effectiveness and hypothesize that 70% of cCBT users will achieve a >50% decline in daily pain ratings.

The investigators will enroll 40 SCD patients at the University of Pittsburgh Medical Center (UPMC) with chronic pain to either CALM-SCD or pain education (eEducation) and follow them for 12 months. Implementation of routine stress/pain screening in the UPMC Adult Sickle Cell Clinic allows investigators to identify patients with SCD who have chronic pain as indicated by self-report "I have had pain nearly every day for at least 3 months" or have been prescribed long-acting opioids for pain.

Following confirmation of protocol-eligibility and informed consent, investigators will provide all patients with a large-screen smartphone (unless the patient owns their own compatible large-screen smartphone) with a symptoms diary app, and GPS tracking features pre-installed; this will allow investigators to track pain and mood as well as any opioid or non-opioid pain treatments used by patients, and steps traveled.

Patients enrolled in the CALM-SCD group will complete at least 4 1-hour cCBT sessions over 3 months using their personal or study-provided smartphone. Because cCBT programs are less effective without a human support component, participants will also be introduced to a care coach (master's level student tech who will receive training in CBT) who will contact them on a weekly basis by phone/text for up to 3 months. The care coach will reinforce CBT materials and encourage engagement. Participants will have continued access to the program after first 3 months, but care coach support will only be available on an as-needed basis.

Patients enrolled in the eEducation group will receive pain education through online modules that they will be asked to complete using their study-provided smartphone. Each module includes learning tasks, a reading assignment, and a short quiz based on material. The education group will receive care coach contact on the same schedule as the cCBT group. The care coach will provide supportive therapy and encouragement to complete modules and apply the lessons to their daily life.

Patients who are not eligible or who are not randomized into one of the intervention arms of this study will serve as a comparison group to ensure we are treating a representative sample of patients. Further, patients who were eligible but were not randomized into one of the intervention arms will serve as a usual care control group.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must be 18 years of age or older, have a documented diagnosis of SCD (HgbSS, HgbSC, SB+Thal, or SBoThal), receive routine care at the UPMC Sickle Cell Clinic, and self-report chronic pain or have been prescribed long-acting opioids for pain.

Exclusion Criteria:

* Unable to provide informed consent due to low literacy or cognitive difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of cognitive behavioral therapy trial for participants | 6 months
  Number of cCBT sessions completed
Feasibility of recruitment and enrollment into cognitive behavioral therapy trial | 3-6 months of open enrollment
  Number of patients enrolled / number of patients screened and approached

SECONDARY OUTCOMES:
Pain intensity | 1, 3, 6, and 12 months
  Average change in 0-10 VAS pain intensity over course of study
Pain interference | 1, 3, 6, and 12 months
  PROMIS Pain Interference
Depressive symptoms | 1, 3, 6, and 12 months
  PHQ-9 depression measure
Anxiety symptoms | 1, 3, 6, and 12 months
  GAD-7 anxiety scale
Pain Catastrophizing Scale | 1, 3, 6, and 12 months
  Pain Catastrophizing
Sickle Cell Self-efficacy Scale | 1, 3, 6, and 12 months
  Self-efficacy
ASCQ-Me | 1, 3, 6, and 12 months
  Quality of life measures

OTHER OUTCOMES:
Activity space | 6 months
  GPS activity tracking on the smartphone

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jonassaint, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
A public-use data set (PUD) will be available through our study website. The PUD will be a cleaned, de-identified copy that includes all enrolled participants. Sensitive, identifying, unreliable, or invalid data will be excluded.
  Researchers may request a copy of the PUD electronically from the Clinical Research Services at the University of Pittsburgh, conditional upon receiving IRB approval for a research proposal from their home institution.